CLINICAL TRIAL: NCT06591481
Title: Retrospective Case-control Study for the Development of an Artificial Intelligence (AI)-Based Tool of Lesion Detection Based on Magnetic Resonance Imaging (MRI) and Clinical Variables for Early Diagnosis of Axial Spondyloarthritis (axSpA)
Brief Title: Retrospective Case-Control Study for Developing an Artificial Intelligence (AI) Tool for Lesion Detection Using Magnetic Resonance Imaging (MRI) and Clinical Variables for Early Diagnosis of Axial Spondyloarthritis (axSpA)
Acronym: InnovaDetect
Status: Completed | Type: Observational
Sponsor: Ángel Alberich Bayarri (Industry)
Responsible Party: Sponsor-Investigator, Ángel Alberich Bayarri, CEO and co-founder of Quibim, Quibim
Organization: Quibim (Industry)
Other Study IDs: axSpA-patients-stratification
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondyloarthritis (AxSpA)
Keywords: Artificial Intelligence; AI; lesion detection; axial Spondyloarthritis; axSpA; MRI; Magnetic Resonance; medical imaging; tool; algorithm; diagnosis; early
MeSH Terms: conditions — Axial Spondyloarthritis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active axSpA patients: Participants diagnosed with axSpA (according to ASAS criteria for axSpA) showing active lesions in their MRI exams.
- Control: This group is composed by: 1) Participants with buttock or low back pain that not fulfil ASAS criteria for axSpA and 2) axSpA patients that do not show active lesions in their MRI exams.

SUMMARY:
The goal of this observational study is to develop and validate an Artificial Intelligence (AI) tool that allows the lesion detection and early diagnosis of axial spondyloarthritis (axSpA) based on Magnetic Resonance Imaging (MRI).

This study will gather MRI scans from axSpA patients and a control group of participants.

DETAILED DESCRIPTION:
BACKGROUND

The spondyloarthritis (SpA) are a group of chronic inflammatory diseases of autoimmune nature that share common clinical and genetic features, including an association with HLA-B27 antigen. They are among the most common rheumatic diseases with a prevalence of 0.01-2,5%. All of these conditions make the patients to move on a chronic disabling disease.

Patients with SpA can be classified based on their clinical presentation into either predominantly axial SpA (axSpA) or predominantly peripheral SpA. Axial SpA is characterized by primary involvement of the sacroiliac joints (SIJs) and/or the spine, leaading to substantial pain and disability. Until recently, the diagnosis of axSpA relied on detecting of structural changes evocative of sacroiliitis in the SIJs using plain radiography.

The introduction of Magnetic resonance imaging (MRI) for evaluating the SIJs has significantly advanced the recognition of axSpA. MRI can detect early inflammatory processes even in patients who do not yet have structural lesions. Besides, MRI has shown superiority over radiography in detecting structural changes in the SIJs. However, the definition of a "positive MRI" in SpA remains controversial, as both sensitivity and specificity have their limitations. Early diagnosis of SpA has become increasingly important, as treatments are now available, and MRI is emerging as the preferred choice for early diagnosis. A number of randomized controlled trials of anti-tumour necrosis factor agents in ankylosing spondylitis have demonstrated regression of inflammatory lesions in the spine by MRI. Moreover, the role of MRI in the early diagnosis of SpA has become better established, and imaging features of active sacroiliitis by MRI have been defined for axSpA diagnosis.

RATIONALE OF THE STUDY

Despite the current advances in medical imaging and ongoing efforts to improve the classification criteria for axSpA, a high proportion of axSpA patients remain under-diagnosed, leading to delays in diagnosis that can result in a poor prognosis. The volume of unstructured data coming from medical imaging contributes to diagnostic delays. The integration of AI and machine learning technologies in medicine for processing large datasets has led to faster and more accurate analysis, identification of real-world evidence gaps, and the agile generation of evidence to address healthcare providers' and healthcare systems' needs.

This study aims to develop an AI diagnostic tool that combines quantitative MRI data with clinical information to aid in the early diagnosis of axSpA.

OBJECTIVES

Primary objective: To create an AI tool that allows the early diagnosis of axSpA and lesion detection based on MRI.

Secondary objective: Clinical validation of the AI module.

Exploratory objective:

* Automated characterization of lesions (oedema, erosion, fat metaplasia and ankylosing) based on texture quantification and radiomics and deep features analysis.
* Determination of normative values for texture imaging biomarker on the SIJs.

SAMPLE DESCRIPTION

The dataset will consist of 900 MRIs, collected retrospectively. MRI exams will be sourced from patients with active axSpA and from those with inactive or no axSpA (control group). The control-to-case ratio will be set at 40/60, allowing the algorithm to learn from both subsets without favoring one group over the other. Since AI can more easily characterize normality than pathology, the proportion of non-axSpA and normal MRIs can be lower (approximately 40%) compared to the 60% allocated to axSpA MRIs. Among the active axSpA group, the distribution of MRIs across classification categories (oedema, ankylosing, erosion, and fat metaplasia) should be as balanced as possible, ideally with 25% assigned to each category. Each MRI does not necessarily come from a different patient, as they may represent different time points for the same individual.

ANALYSIS PLAN

1. Image Quality Control.

   All the images received from sites will be checked by imaging technicians to guarantee the homogeneity of the data
2. Centralized Image Interpretation.

   A centralized radiological review of the MRI images will be conducted by senior MSK expert radiologists. Each case will be evaluated by two radiologists. If there is a disagreement between the two, a third radiologist will review the case.

   The radiologists will classify the MRIs into the study's various classes and cohorts based on the ASAS criteria for defining active sacroiliitis on MRI for the classification of axial spondyloarthritis. All radiologists involved in the project will receive training to detect lesions according to the ASAS criteria, and this training will be documented and stored in the study's repository.
3. Annotation process.

   The imaging technicians will delineate the lesions detected by the MSK expert radiologists to generate a 3D volume. This will be then reviewed by the MSK expert radiologist.
4. Imaging Biomarkers Extraction.

   To obtain further information of the lesions labeled, a texture analysis will be performed to quantify several features related to the heterogeneity of the tissue that can be considered as an indicator of the pathological process. The radiomic panel will be based on the following features:
   * Structural or shape features: Descriptive of the geometric properties of the image. Examples of these features are volume, maximum orthogonal diameter, maximum surface area, compactness, fractal dimension or sphericity of a lesion.
   * Statistical characteristics are those that are inferred by statistical relationships. They can be in turn:

     * First-order or distributional: They provide information on the frequency of individual voxel values without taking into consideration their spatial relationships. This distribution is presented in the form of histograms, which report the mean, median, maximum and minimum in the intensities of the voxels, but also on the asymmetry, kurtosis, uniformity or entropy of the distribution.
     * Second order or texture: They reflect the relationships between neighboring voxels, allowing to obtain a spatial arrangement of their intensities, thus giving an idea about the architecture and heterogeneity of the studied tissue. These relationships are obtained by means of statistical analyses, such as cooccurrence matrices, which measure the probability that two neighboring voxels have the same signal intensity.
     * Higher order: These are combinations of features obtained by complex statistical analysis, such as fractal analysis, on images to which filters or mathematical transformations have been applied to maximize or minimize patterns, remove noise, or highlight certain details.
   * Deep features: These are properties obtained by analyzing images with convolutional neural networks (CNN) or other deep learning algorithms. These algorithms are trained to be able, in an image, to automatically determine and select those features or sets of classifying features, without the need of human intervention.
5. AI Module Development.

Using the MRIs collected together with the imaging biomarkers and other clinical information available, the data scientists will create an AI-based model that will provide a probability score of axSpA for each subject.

To create the AI module, the database will be divided in three non-balanced sub datasets (training, validation and test). The bigger dataset of images will be used for training the module. After the training phase, the validation database will be used to check if the classification is well done or the model should be trained again.

Training: Set of cases used to fit the model during the training process. These will be the cases the model will use to tune its weights, i.e. the cases that the model will use to "learn".

Validation: Set of cases used to evaluate the model during the training process, therefore, are not used to tune the model weights. This dataset is used for three main purposes:

* Hyperparameters tuning.
* Overfitting detection: During the training process, after each training iteration (epoch), the model is evaluated over both the training and validation datasets.
* Selection of the "best" model during the training process, this means that the weights from the training iteration in which the best validation metrics are obtained are stored.

Test: A separate set, not used for training or validation, will be used for the final model evaluation.

In this study, MRI exams will be obtained from various scanners and institutions. Therefore, the acquisition protocols and reconstruction techniques may vary between scanners. To address this, preprocessing techniques will be applied to standardise the images across different scanners.

ELIGIBILITY:
Inclusion Criteria for Active axSpA patients group:

* Fulfillment of the ASAS criteria for axSpA (i.e. MRI and/or clinical arm, Rudwaleit M, et al., Ann Rheum Dis. 2009 Oct;68(10):1520-7).
* axSpA diagnosis according to the physician.
* Fulfillment of the following MRI criteria (a-c must be fulfilled):
* a) Availability of MRI images of the sacroiliac joint (SIJ) including T1- weighted and STIR and/or T2 Fat-Sat (FS) sequences in coronal-oblique planes.
* b) Fulfillment of ASAS criteria for positive MRI:
* b.1)Bone marrow oedema (BMO) on a T2-weighted sequence sensitive for free water (such as short tau inversion recovery [STIR] or T2FS) or bone marrow contrast enhancement on a T1-weighted sequence (such as T1FS post-gadolinium).
* b.2) Inflammation must be clearly present and located in a typical anatomical area (subchondral bone).
* b.3) MRI appearance must be highly suggestive of SpA.
* b.4) Other findings can be present but are not required for a positive MRI (erosion and/or fat metaplasia and/or ankylosis).
* b.5) Fulfillment of ASAS criteria for positive MRI.
* c) MRI expert opinion of having axial SpA.

Inclusion Criteria for Control group:

* Buttock and/or low back pain due to known trauma, stress, disc herniation with an MRI of SIJ showing absence of bone marrow edema, fatty infiltration and bone erosions and not fulfilling ASAS axSpA classification criteria.
* Availability of MRI images of SIJ including T1-weighted and STIR and/or T2 Fat-Sat sequences in coronal-oblique planes.

Exclusion Criteria:

* Another known pathology in the SIJ which may influence the MRI interpretation.
* Unreadable MRI images or with insufficient diagnostic quality.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants come from 4 different countries within the EMEA region (Spain, United Arab Emirates, Jordan and Saudi Arabia)
Sampling Method: Non-Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2023-02-19 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | From diagnosis until sample completion (an average of 2 years)
  The metric used for parameter optimization and model selection will be the area under the curve (AUC) for balanced dataset.
F1 score | From diagnosis until sample completion (an average of 2 years)
  In case of unbalanced dataset, F1 score will be used for parameter optimization and model selection.
Balanced accuracy | From diagnosis until sample completion (an average of 2 years)
Matthews correlation coefficient | From diagnosis until sample completion (an average of 2 years)
Sensitivity | From diagnosis until sample completion (an average of 2 years)
Specificity | From diagnosis until sample completion (an average of 2 years)

CONTACTS AND LOCATIONS:
Locations (7):
- Royal Medical Services, Amman, Jordan
- King Saud Medical City, Riyadh, Saudi Arabia
- General University Hospital of Valencia, Valencia, Valencia, Spain
- United Arab Emirates (4):
  - Tawam hospital (SEHA), Al Ain City, Al Maqam
  - Cleveland Clinic Abu Dhabi, Abu Dhabi
  - YAS Clinic, Abu Dhabi
  - Emirates Health Services (EHS), Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudwaleit M, Jurik AG, Hermann KG, Landewe R, van der Heijde D, Baraliakos X, Marzo-Ortega H, Ostergaard M, Braun J, Sieper J. Defining active sacroiliitis on magnetic resonance imaging (MRI) for classification of axial spondyloarthritis: a consensual approach by the ASAS/OMERACT MRI group. Ann Rheum Dis. 2009 Oct;68(10):1520-7. doi: 10.1136/ard.2009.110767. Epub 2009 May 18. PMID 19454404
- [Background] Lambert RG, Bakker PA, van der Heijde D, Weber U, Rudwaleit M, Hermann KG, Sieper J, Baraliakos X, Bennett A, Braun J, Burgos-Vargas R, Dougados M, Pedersen SJ, Jurik AG, Maksymowych WP, Marzo-Ortega H, Ostergaard M, Poddubnyy D, Reijnierse M, van den Bosch F, van der Horst-Bruinsma I, Landewe R. Defining active sacroiliitis on MRI for classification of axial spondyloarthritis: update by the ASAS MRI working group. Ann Rheum Dis. 2016 Nov;75(11):1958-1963. doi: 10.1136/annrheumdis-2015-208642. Epub 2016 Jan 14. PMID 26768408
- [Background] Huang Y, Chen Y, Liu T, Lin S, Yin G, Xie Q. Impact of tumor necrosis factor alpha inhibitors on MRI inflammation in axial spondyloarthritis assessed by Spondyloarthritis Research Consortium Canada score: A meta-analysis. PLoS One. 2020 Dec 31;15(12):e0244788. doi: 10.1371/journal.pone.0244788. eCollection 2020. PMID 33382842
- [Background] Lukas C, Cyteval C, Dougados M, Weber U. MRI for diagnosis of axial spondyloarthritis: major advance with critical limitations 'Not everything that glisters is gold (standard)'. RMD Open. 2018 Jan 12;4(1):e000586. doi: 10.1136/rmdopen-2017-000586. eCollection 2018. PMID 29479474
- [Background] Khmelinskii N, Regel A, Baraliakos X. The Role of Imaging in Diagnosing Axial Spondyloarthritis. Front Med (Lausanne). 2018 Apr 17;5:106. doi: 10.3389/fmed.2018.00106. eCollection 2018. PMID 29719835
- [Background] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Akkoc N, Brandt J, Chou CT, Dougados M, Huang F, Gu J, Kirazli Y, Van den Bosch F, Olivieri I, Roussou E, Scarpato S, Sorensen IJ, Valle-Onate R, Weber U, Wei J, Sieper J. The Assessment of SpondyloArthritis International Society classification criteria for peripheral spondyloarthritis and for spondyloarthritis in general. Ann Rheum Dis. 2011 Jan;70(1):25-31. doi: 10.1136/ard.2010.133645. Epub 2010 Nov 24. PMID 21109520
- [Background] Stolwijk C, Boonen A, van Tubergen A, Reveille JD. Epidemiology of spondyloarthritis. Rheum Dis Clin North Am. 2012 Aug;38(3):441-76. doi: 10.1016/j.rdc.2012.09.003. PMID 23083748